CLINICAL TRIAL: NCT02458391
Title: Therapeutic Quantity of Complete Decongestive Therapy in Breast Cancer-Related Lymphedema: A Double Blinded Randomized Control Trial
Brief Title: Complete Decongestive Therapy in Breast Cancer-Related Lymphedema
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants available
Sponsor: University of Indianapolis (Other)
Collaborators: Novacare (Unknown); Midwestern University (Other)
Responsible Party: Principal Investigator, Katie M. Polo, MHS, OTR/L, CLT-LANA, Sponsor Investigator, University of Indianapolis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UIndianapolis
Record Dates: First submitted 2014-11-17; First posted 2015-06-01 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Lymphedema of Upper Limb
Keywords: Breast Cancer; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment 2x/wk (Experimental): Participants will receive standard of care complete decongestive therapy 2x/wk for 4 weeks.
  Interventions: Other: Standard of care complete decongestive therapy
- Treatment 4x/wk (Experimental): Participants will receive standard of care complete decongestive therapy 4x/wk for 4 weeks.
  Interventions: Other: Standard of care complete decongestive therapy

INTERVENTIONS:
Other: Standard of care complete decongestive therapy — Participants will receive standard of care complete decongestive therapy consisting of meticulous skin and nail care, manual lymphatic drainage, compression bandaging, remedial exercises and self-care training.

SUMMARY:
The purpose of this study is to investigate which number of lymphedema therapy treatments/week best reduces upper extremity swelling, increased arm function, and reduces the most lymphedema symptoms.

DETAILED DESCRIPTION:
Complete Decongestive Therapy (CDT) is the "gold standard" in lymphedema care and has been found to be efficacious in numerous studies. These studies have varying treatment protocols of intensive phase I CDT with dosing ranging from 2x/wk for a mean of 7.5 wks to 6x/wk until a plateau in arm volumes were achieved. This variability in research does not lend itself to recommendations of evidence-based protocol use of CDT in an outpatient setting.

Although CDT is backed by efficacy studies, the daily dosing given to patients is based on anecdotal rather than evidence-based practice. Because the traditional protocol was developed from "longstanding experience," research is necessary to determine the best dosing of the intensive phase of CDT. The purpose of this study is to investigate what level of dosing in the intensive CDT phase promotes best volume reduction and increased upper extremity function in the breast cancer-related lymphedema patient population. This particular study will answer: What dosing produces best volumetric reduction and upper extremity function in the intensive phase of complete decongestive therapy for outpatients with breast cancer-related lymphedema 2x/wk for 4wks or 4x/wk for 4 wks?

ELIGIBILITY:
Inclusion Criteria:

1. Have active unilateral breast cancer-related lymphedema
2. Medically stable
3. Have not participated in lymphedema therapy the past 3 months
4. An affected limb volume measurement of >10% excess volume
5. Ages 18-95 years old

   * Patients undergoing any medical treatment for their breast cancer diagnosis will be included in this study.
   * Patients with any stage breast cancer will be included in this study.
   * Patients with a prior diagnosis of breast cancer, other cancer will be included in this study. There is no minimum time requirement that has prolapsed between their diagnosis and this study.

All subjects must have given signed, informed consent prior to registration on study.

Exclusion Criteria:

1. Prophylactic treatment indicated
2. A presence of upper extremity wounds present
3. Active signs of infection or deep vein thrombosis (DVT)
4. Bilateral lymphedema present
5. Evidence of contraindications to CDT: uncontrolled hypertension, heart disease including congestive heart failure, and renal insufficiency
6. Severe lymphedema present as defined by > 30% increase in limb volume

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in impairments in function, activity limitations, and participation restrictions | At first treatment appointment (roughly week 1), after 4 weeks of treatment, at discharge (roughly after 8 weeks), and at a 4 week follow-up session after discharge (up to 12 weeks)
  A questionnaire looking at impairments in function, activity limitations, and participation restrictions consists of 29 questions divided into five domains: physical function, mental function, household activities, mobility activities, and life and social activities.
Changes from baseline in symptoms associated with lymphedema | At first treatment appointment (week 1), after 4 weeks of treatment, at discharge (roughly after 8 weeks), and at a 4 week follow-up session after discharge (up to 12 weeks)
  This outcome measure will assess the presence of symptoms associated with lymphedema.

SECONDARY OUTCOMES:
Changes from baseline in lymphedema volume | At first treatment appointment (week 1), after 4 weeks of treatment, at discharge (roughly after 8 weeks), and at a 4 week follow-up session after discharge (up to 12 weeks)
  Circumferential measurements by tape measure calculated into volume percentage

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rundquist, PhD, PT, Principal Investigator — University of Indianapolis

REFERENCES:
- [Result] Fu, M.R., Hu, S. Cleland, C.M. Kang, Y. (June, 29, 2012). Measuring lymphedema symptom burdens: A psychometric study. The Multinational Association of Supportive Care in Cancer's annual meeting (MASCC/ISOO): 2012 International Symposium on Supportive Care in Cancer in New York City on June 28-30, 2012.
- [Result] Mayrovitz HN, Macdonald J, Davey S, Olson K, Washington E. Measurement decisions for clinical assessment of limb volume changes in patients with bilateral and unilateral limb edema. Phys Ther. 2007 Oct;87(10):1362-8. doi: 10.2522/ptj.20060382. Epub 2007 Aug 7. PMID 17684090
- [Result] Taylor R, Jayasinghe UW, Koelmeyer L, Ung O, Boyages J. Reliability and validity of arm volume measurements for assessment of lymphedema. Phys Ther. 2006 Feb;86(2):205-14. PMID 16445334
- [Result] Devoogdt N, Van Kampen M, Geraerts I, Coremans T, Christiaens MR. Lymphoedema Functioning, Disability and Health questionnaire (Lymph-ICF): reliability and validity. Phys Ther. 2011 Jun;91(6):944-57. doi: 10.2522/ptj.20100087. Epub 2011 Apr 14. PMID 21493748